CLINICAL TRIAL: NCT07012447
Title: Evaluating the Efficacy of Venetoclax Combined With Azacitidine Induction Therapy of Early T-cell Precursor-like Acute Lymphoblastic Leukemia and T-ALL With Myeloid Mutations
Brief Title: Venetoclax + Azacytidine for Newly Diagnosed ETP-like ALL and T-ALL With Myeloid Mutations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: yuejun Liu (Other)
Responsible Party: Sponsor-Investigator, yuejun Liu, Physician, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ-ETP01
Record Dates: First submitted 2025-04-21; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Early T Acute Lymphoblastic Leukemia; T-Acute Lymphoblastic Leukemia; Mixed Phenotype Acute Leukemia, T/Myeloid, Nos
Keywords: Adverse risk; newly diagnosed; induction therapy
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Pyloric Stenosis, Hypertrophic | interventions — venetoclax; Azacitidine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational ( venetoclax, azacytidine) (Experimental): Two cycles induction as venetoclax (oral, 100 mg D1, 200 mg D2, 400 mg D3-28) and azacitidine (75 mg/m² SC D1-7); Consolidation: For fit patients, if those with MRD (Minimal Residual Disease) are negative or refuse to undergo allo-HSCT (Hematopoietic stem-cell transplantation), intermediate-dose (2g/m² q12h, days 1-3) cytarabine-based therapy is administered for 3-4 cycles; if patients are MRD-positive, they undergo allo-HSCT.
  For unfit patients, each venetoclax combined with azacitidine treatment cycle is anticipated to be 28 days in length until progression of disease, although cycle delays may occur due to delayed blood count recovery.
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: Cytarabine

INTERVENTIONS:
Drug: Venetoclax — Orally by mouth
  Other Names: Venclexta
Drug: Azacitidine — Subcutaneous injection
Drug: Cytarabine — Intravenous infusion
  Other Names: Ara-C

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of venetoclax combined with azacitidine in treating newly diagnosed early T-cell precursor (ETP)-like acute lymphoblastic leukemia (ALL), T-ALL with myeloid mutations, or T/myeloid mixed-phenotype acute leukemia (T/My-MPAL).

Participant population: Patients aged ≥14 years diagnosed with ETP-like leukemia, T-ALL with myeloid mutations, or T/My-MPAL, regardless of sex/gender.

The main question it aims to answer: Does venetoclax plus azacitidine achieve a significantly higher overall response rate (ORR: CR + CRi) compared to historical controls (54% vs. 90%) after two induction cycles?

Comparison group: Researchers will compare ORR outcomes to historical data from conventional chemotherapy regimens to assess treatment superiority.

Participants will:

* Receive two 28-day cycles of venetoclax (oral, 100 mg D1, 200 mg D2, 400 mg D3-28) and azacitidine (75 mg/m²/day SC, D1-7).
* Undergo serial bone marrow biopsies, blood tests, and imaging (e.g., PET-CT) for response assessment.
* Follow dose adjustment protocols for toxicity management (e.g., neutropenia, thrombocytopenia).

DETAILED DESCRIPTION:
This study addresses the unmet need for effective therapies in high-risk T-ALL subtypes, including ETP-like leukemia and T/My-MPAL, which exhibit myeloid-like genetic profiles (e.g., FLT3, DNMT3A, RUNX1 mutations) and poor outcomes under conventional chemotherapy (5-year OS <40%). Preclinical and pilot clinical data demonstrate that venetoclax, a BCL-2 inhibitor, synergizes with azacitidine, a hypomethylating agent, to induce apoptosis in leukemia stem cells by targeting oxidative phosphorylation and epigenetic dysregulation. Building on a pilot study, this Phase II trial employs a single-arm design to validate efficacy in a larger cohort.

Patients receive two induction cycles of venetoclax (oral, 100 mg D1, 200 mg D2, 400 mg D3-28) and azacitidine (75 mg/m² SC D1-7), with response assessed via bone marrow morphology, flow cytometry, and molecular testing (Days 22-35).

Early Efficacy Evaluation: After the first induction cycle (Days 22-35), response is assessed via bone marrow morphology, flow cytometry, and molecular profiling.

Stopping Criteria:

Patients failing to achieve at least partial remission (PR) after Cycle 1 will be withdrawn from the study.

Patients failing to achieve CR or CRi at the end of Cycle 2 will also discontinue study treatment.

Consolidation strategies include allo-HSCT or high dose cytarabine (HiDAC) for fit patients or maintenance therapy for unfit individuals.

Rigorous safety monitoring follows NCI-CTCAE v5.0 criteria, with dose adjustments for hematologic/non-hematologic toxicities.

Statistical analysis includes intent-to-treat and per-protocol populations, with ORR analyzed via exact binomial tests and survival endpoints via Kaplan-Meier/Cox regression. The study integrates translational biomarkers (e.g., BCL-2 expression, mutational profiling) to identify predictors of response, aiming to establish a novel, mechanism-driven regimen for these aggressive leukemias.

ELIGIBILITY:
Inclusion Criteria:

1. No gender restrictions
2. Age ≥ 14 years
3. Confirmed diagnosis of one of the following:

   ETP-like leukemia (CD7⁺, CD1a-, CD8-, with CD5 expression stratified as ETP-ALL ≤75% or Near-ETP-ALL >75%) T-cell acute lymphoblastic leukemia (T-ALL) with myeloid mutations (including FLT3, DNMT3A, STAG2, IDH1/2, RUNX1, EZH2, WT1, ASXL1/2, SF3B1, TET2, BCOR, BCORL1, and MLL-PTD) T/myeloid mixed phenotype acute leukemia (T/My-MPAL) (with concurrent T-lineage and myeloid markers, e.g., cCD3⁺/mCD3⁺, CD7⁺, MPO⁺)
4. Newly diagnosed patients without prior induction therapy Limited prior therapy allowed: hydroxyurea, dexamethasone, or low-dose cytarabine/venetoclax (cumulative dose <0.5g), and leukocytapheresis
5. Expected survival time ≥ 3 months
6. Liver function: total bilirubin ≤ 2× ULN; ALT/AST ≤ 3× ULN (or ≤ 5× ULN if liver infiltration by leukemia is present) ; Renal function: endogenous creatinine clearance ≥ 30 ml/min; Cardiac function: left ventricular ejection fraction > 45%
7. Demonstrated capacity to understand the study and willingness to provide informed consent

Exclusion Criteria:

1. Presence of recurrent genetic abnormalities such as t(8;21), t(15;17), inv(16)/t(16;16) leukemia
2. Prior hypersensitivity to study drugs or compounds of similar chemical structure
3. Active uncontrolled infections as determined by the investigator
4. Active bleeding
5. Recent history (within 1 year) of thrombosis, embolism, or cerebral hemorrhage
6. Pregnancy, breastfeeding, or unwillingness to use contraception in women of childbearing potential
7. Drug addiction or chronic alcoholism that could interfere with trial evaluation
8. Psychiatric disorders or other conditions that would prevent obtaining informed consent or compliance with trial requirements
9. Any condition deemed unsuitable for trial participation by the investigator

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) after two treatment cycles of induction therapy | time from the date of enrollment to 2 cycles of induction before consolidation therapy（100 days）
  Rates of complete remission (CR), and complete remission with incomplete hematologic recovery (CRi)

SECONDARY OUTCOMES:
OS: overall survival | 2 years
  time from the date of enrollment to death from any cause or the last follow-up
LFS：leukemia-free survival | 2 years
  the duration from the date of enrollment to the occurrence of treatment failure, relapse, death from any cause, or the last follow-up.
DOR: duration of remission | 2 years
  Time between the first remission and relapse
AE | Within 60 days after treatment
  Adverse events during the induction treatment.
Volume of infused blood products | Within 60 days
  The volume of infused blood products during the induction treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yue-jun Liu, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- Ethical Committee of the First Affliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No